CLINICAL TRIAL: NCT01050257
Title: A Multicenter Study of the Safety of Oseltamivir Administered Intravenously for the Treatment of Influenza in Patients Aged Greater Than or Equal to 13 Years
Brief Title: A Study of Intravenously Administered Tamiflu (Oseltamivir) in Patients Over 13 Years of Age With Influenza
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NV25118
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Results first posted 2013-11-01 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-08

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Oseltamivir (TAMIFLU®) 100 mg (Experimental): Oseltamivir (TAMIFLU®) 100 mg intravenous (IV) infused over 2 hours, two times a day (every 12 hours) for 5 days. At the discretion of the investigator after 3 days of treatment (6 doses), participants could either continue IV treatment or switch to 75 mg oral oseltamivir twice daily to complete the 5 days of treatment. If necessary, after completing the 5 days of treatment, participants could receive additional treatment with study drug (IV or oral) for up to 5 days.
  Interventions: Drug: Oseltamivir IV; Drug: Oseltamivir Oral
- Oseltamivir (TAMIFLU®) 200 mg (Experimental): Oseltamivir (TAMIFLU®) 200 mg intravenous (IV) infused over 2 hours, two times a day (every 12 hours) for 5 days. At the discretion of the investigator after 3 days of treatment (6 doses), participants could either continue IV treatment or switch to 150 mg oral oseltamivir twice daily for 5 days. If necessary, after completing the 5 days of treatment, participants could receive additional treatment with study drug (IV or oral) for up to 5 days.
  Interventions: Drug: Oseltamivir IV; Drug: Oseltamivir Oral
- Oseltamivir Open Label (Experimental): Moderate/Severe renal impaired participants received open label oseltamivir IV or oseltamivir capsules at reduced doses for 5 days as per protocol. If necessary, after completing the 5 days of treatment, participants could receive additional treatment with study drug as per protocol.
  Interventions: Drug: Oseltamivir IV; Drug: Oseltamivir Oral

INTERVENTIONS:
Drug: Oseltamivir IV — Oseltamivir IV infusions over 2 hours two times a day (every 12 hours) for 5 days for patients with moderate renal impairment. Patients with severe renal impairment received once daily dosing and patients on renal replacement therapy received dose/frequency according to protocol.
  Other Names: TAMIFLU®
Drug: Oseltamivir Oral — Oseltamivir (TAMIFLU®) capsules taken orally for 5 days. Twice daily (every 12 hours) for patients with moderate renal impairment, once daily for patients with severe renal impairment and dose frequency according to protocol for patients on renal replacement therapy.
  Other Names: TAMIFLU®

SUMMARY:
This partially randomized, multi-center parallel-group study will evaluate the safety, pharmacokinetics and the effect on viral load and viral shedding of Tamiflu (Oseltamivir) in patients with influenza. Adult and adolescent patients will be randomized to receive either 100 mg or 200 mg of study drug intravenously every 12 hours. Investigators and patients are blinded to knowledge of the assigned dose of Tamiflu. There is an option to convert to oral Tamiflu after 6 intravenous infusions. The anticipated time on study treatment is 5 days, with an optional treatment extension of a further 5 days, if necessary. There will be a non-randomized, open-label treatment group for patients with moderate/severe renal impairment or renal failure. Intravenous dose levels and frequency will be adjusted appropriately to their renal situation.

ELIGIBILITY:
Inclusion Criteria:

* Adult and adolescent patients, 13 years of age and older
* Diagnosis of influenza
* ≤ 144 hours between the onset of influenza-like illness and first dose of study drug

Non-randomized, open-label treatment group:

* Patients with moderate/severe renal impairment or renal failure with creatinine clearance 10-60 mL/min

Exclusion Criteria:

* Clinical evidence of severe hepatic decompensation at the time of randomization
* Acute ischemia or significant arrhythmia

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2010-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (87):
- United States (50):
  - Birmingham, Alabama
  - Montgomery, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Duarte, California
  - Los Angeles, California
  - San Diego, California
  - Wilmington, Delaware
  - Melbourne, Florida
  - Miami, Florida
  - Pensacola, Florida
  - South Miami, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Maywood, Illinois
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Overland Park, Kansas
  - Wichita, Kansas
  - Madisonville, Kentucky
  - New Orleans, Louisiana
  - Worcester, Massachusetts
  - Detroit, Michigan
  - Kalamazoo, Michigan
  - Duluth, Minnesota
  - Minneapolis, Minnesota
  - Jackson, Mississippi
  - Saint Joseph, Missouri
  - Butte, Montana
  - Grand Island, Nebraska
  - Holmdel, New Jersey
  - New York, New York
  - South Bronx, New York
  - Stony Brook, New York
  - The Bronx, New York
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Youngstown, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Dallas, Texas
  - San Antonio, Texas
  - Norfolk, Virginia
  - Charleston, West Virginia
- Odense C, Denmark
- France (5):
  - Bron
  - Garches
  - La Tronche
  - Paris
  - Tours
- Hungary (13):
  - Budapest
  - Debrecen
  - Eger
  - Győr
  - Gyula
  - Kaposvár
  - Miskolc
  - Nyíregyháza
  - Pécs
  - Szeged
  - Szolnok
  - Szombathely
  - Veszprém
- Italy (5):
  - Genova
  - Milan
  - Monza
  - Pavia
  - Roma
- Lithuania (2):
  - Kaunas
  - Vilnius
- Poland (4):
  - Bialystok
  - Chorzów
  - Radom
  - Warsaw
- Romania (4):
  - Bucharest
  - Constanța
  - Craiova
  - Timișoara
- Spain (3):
  - Elche, Alicante
  - Almería, Almeria
  - Madrid, Madrid

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included a 5 day treatment period and an optional extension. Participants were considered to have completed treatment if they completed the 5-day course of treatment (IV and/or oral).
Period: Overall Study
Arm/Group | Oseltamivir (TAMIFLU®) 100 mg | Oseltamivir (TAMIFLU®) 200 mg | Oseltamivir Open Label
Started | 50 | 53 | 15
Received Treatment | 49 | 50 | 14
Safety Population: Actual Dose Received | 48 | 51 (One participant randomized to 100 mg actually received the 200 mg doses.) | 14
Intent-to-treat Infected Confirmed | 30 | 32 | 10
Switched to Oral Treatment | 28 | 31 | 3
Completed | 39 (Completed 5 days of treatment either IV or Oral) | 40 | 8
Not Completed | 11 | 13 | 7
Not completed — Adverse Event | 4 | 4 | 2
Not completed — Admin/Other (did not switch to oral) | 6 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 3 | 0
Not completed — No reason specified | 0 | 0 | 2
Not completed — Refused treatment/ Did not Cooperate | 1 | 1 | 0
Not completed — Violation criteria | 0 | 1 | 0
Not completed — Failure to return | 0 | 2 | 0
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Demographics are based on the all enrolled patients population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oseltamivir (TAMIFLU®) 100 mg | Oseltamivir (TAMIFLU®) 200 mg | Oseltamivir Open Label | Total
Number analyzed (Participants) | 50 | 53 | 15 | 118
Age Continuous [Mean (Standard Deviation); unit: years] | 44.8 (16.68) | 44.3 (18.09) | 66.9 (18.28) | 47.4 (18.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 8 | 60
  Male | 25 | 26 | 7 | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events(SAEs, AEs Leading to Withdrawal, and Death
Description: Safety was assessed by adverse events (AEs) as measured by the collection of AEs, vital signs, electrocardiograms and laboratory parameters. An AE was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study were reported as adverse events. A serious adverse event is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
  On treatment = AEs that started between the day of first dose and within 2 days after the last dose. Off treatment = AEs that started more than 2 days after the last dose of study drug.
Time Frame: Up to 30 days
Population: Safety population included all participants who received treatment and had at least one post-treatment safety assessment. One patient in the 100 mg group actually received 200 mg and is included in the 200 mg group for safety.
Measure: Number; unit: Partipants
Arm/Group | Oseltamivir (TAMIFLU®) 100 mg | Oseltamivir (TAMIFLU®) 200 mg | Oseltamivir Open Label
Number analyzed (Participants) | 48 | 51 | 14
Partipants
  Death | 1 | 1 | 3
  AEs on treatment: IV dose | 24 | 27 | 11
  AEs on treatment: Oral dose | 10 | 9 | 4
  AEs off treatment | 13 | 13 | 5
  SAEs on treatment: IV dose | 3 | 4 | 2
  SAEs on treatment: Oral dose | 2 | 0 | 2
  SAEs off treatment | 5 | 1 | 3
  AEs leading to withdrawal on treatment: IV dosing | 3 | 3 | 2
  AEs leading to withdrawal on treatment: Oral dose | 1 | 1 | 1
  AEs leading to withdrawal off treatment | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics
Time Frame: Days 1, 3
Reporting Status: Not Posted, anticipated posting 2013-12

3. Secondary Outcome: Percentage of Participants With Viral Shedding by Culture or RT-PCR
Description: Nasal and throat swabs were collected on Days 1, 4, 6, 11, 15, and 30 and were sent to a central laboratory for analysis. The presence of viral shedding was determined by a positive culture [log10 median tissue culture infective dose (TCID50) > 0.5) or detection by RT-PCR (log 10 copies/mL).
Time Frame: Days 1, 4, 6, 11, 15 and 30
Population: Intent-to-Treat Infected population included all treated participants who had confirmed influenza infection by culture or RT-PCR.
Measure: Number; unit: Percentage of participants
Arm/Group | Oseltamivir (TAMIFLU®) 100 mg | Oseltamivir (TAMIFLU®) 200 mg | Oseltamivir Open Label
Number analyzed (Participants) | 30 | 32 | 10
Percentage of participants
  Day 1 (n=29, 30, 10) | 90 | 97 | 90
  Day 4 (n=28, 28, 10) | 64 | 75 | 60
  Day 6 (n=22, 28, 8) | 41 | 36 | 63
  Day 11 (n=22, 26, 8) | 9 | 15 | 13
  Day 15 (n=17, 24, 7) | 0 | 8 | 14
  Day 30 (n=22, 28, 6) | 5 | 4 | 0

4. Secondary Outcome: Percentage of Participants With Viral Shedding by Culture
Description: Nasal and throat swabs were collected on Days 1, 4, 6, 11, 15, and 30 and were sent to a central laboratory for analysis. The presence of viral shedding was determined by a positive culture=log10 median tissue culture infective dose (TCID50) > 0.5.
Time Frame: Days 1, 4, 6, 11, 15, 30
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Oseltamivir (TAMIFLU®) 100 mg | Oseltamivir (TAMIFLU®) 200 mg | Oseltamivir Open Label
Number analyzed (Participants) | 30 | 32 | 10
Percentage of participants
  Day 1 (n=29, 30, 10) | 76 | 80 | 90
  Day 4 (n=28, 28, 10) | 14 | 29 | 30
  Day 6 (n=22, 28, 8) | 5 | 0 | 0
  Day 11 (n=22, 26, 8) | 0 | 4 | 0
  Day 15 (n=17, 24, 7) | 0 | 4 | 14
  Day 30 (n=22, 28, 6) | 5 | 4 | 0

5. Secondary Outcome: Percentage of Participants With Viral Shedding by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR)
Description: Nasal and throat swabs were collected on Days 1, 4, 6, 11, 15, and 30 and were sent to a central laboratory for analysis. The presence of viral shedding was determined by detection by RT-PCR (log 10 copies/mL).
Time Frame: Days 1, 4, 6, 11, 15 and 30
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Oseltamivir (TAMIFLU®) 100 mg | Oseltamivir (TAMIFLU®) 200 mg | Oseltamivir Open Label
Number analyzed (Participants) | 30 | 32 | 10
Percentage of participants
  Day 1 (n=29, 30, 10) | 86 | 93 | 90
  Day 4 (n=28, 28, 10) | 64 | 71 | 60
  Day 6 (n=22, 28, 8) | 41 | 36 | 63
  Day 11 (n=22, 26, 8) | 9 | 12 | 13
  Day 15 (n=17, 24, 7) | 0 | 4 | 0
  Day 30 (n=22, 28, 6) | 5 | 4 | 0

6. Secondary Outcome: Change From Baseline in Influenza Titer by Culture at Day 4
Description: Nasal and throat swabs collected at Baseline and Day 4 were sent to a laboratory for analysis. Viral influenza titer (amount of virus present) was determined by culture. A log 10 median tissue culture infective dose (TCID50) > 0.5= Positive culture. A negative change from Baseline indicated improvement (less virus present).
Time Frame: Baseline, Day 4
Population: Participants from the Intent-to-treat Influenza Infected population with data available for analysis. Only participants with positive influenza results are included.
Measure: Mean (Standard Deviation); unit: log10 TCID50
Arm/Group | Oseltamivir (TAMIFLU®) 100 mg | Oseltamivir (TAMIFLU®) 200 mg | Oseltamivir Open Label
Number analyzed (Participants) | 4 | 8 | 3
log10 TCID50 | -1.38 (1.920) | -2.19 (1.186) | -3.00 (0.750)

7. Secondary Outcome: Change From Baseline in Influenza Titer by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) at Day 4
Description: Nasal and throat swabs were collected at Baseline and Day 4 and were sent to a central laboratory for analysis. Influenza Viral titers (amount of virus present) were determined by RT-PCR for Flu A and Flu B and were reported in log 10 copies/milliliter (mL). A negative change from Baseline indicated improvement (less virus present).
Time Frame: Baseline, Day 4
Population: Participants from the Intent-to-Treat Infected population with data available for analysis. Only participants with positive influenza results are included.
Measure: Mean (Standard Deviation); unit: log 10 copies/mL
Arm/Group | Oseltamivir (TAMIFLU®) 100 mg | Oseltamivir (TAMIFLU®) 200 mg | Oseltamivir Open Label
Number analyzed (Participants) | 30 | 32 | 10
log 10 copies/mL
  Flu A (n=14, 14, 5) | -1.04 (1.412) | -1.30 (0.883) | -1.53 (0.930)
  Flu B (n=3, 5, 1) | -0.70 (1.459) | -1.51 (0.262) | -2.27 (NA) — Unable to calculate standard deviation, data available for only 1 patient.

8. Secondary Outcome: Percentage of Participants Who Had a Fever During the Study
Description: Fever was defined as a temperature of ≥ 37.8 C (degrees Celcius).
Time Frame: Baseline and Hours 12, 24, 36, 48, 60, 72, 84, 96 and 108
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Oseltamivir (TAMIFLU®) 100 mg | Oseltamivir (TAMIFLU®) 200 mg | Oseltamivir Open Label
Number analyzed (Participants) | 30 | 32 | 10
Percentage of participants
  Baseline | 23 | 19 | 20
  Hour 12 | 7 | 9 | 10
  Hour 24 | 7 | 0 | 0
  Hour 36 | 3 | 3 | 20
  Hour 48 | 3 | 6 | 0
  Hour 60 | 0 | 6 | 0
  Hour 72 | 0 | 3 | 0
  Hour 84 | 0 | 0 | 0
  Hour 96 | 0 | 3 | 0
  Hour 108 | 0 | 0 | 0

9. Secondary Outcome: Time to Resolution of Fever for Participants Who Had a Fever at Baseline
Description: Fever was defined as a temperature of ≥ 37.8 C (degrees Celsius). Resolution of fever was a temperature ≤ 37.2 for at least 21.5 hours.
Time Frame: Baseline, Up to 30 Days
Population: Participants from the Intent-to-Treat Infected population, all treated participants with confirmed influenza infection by culture or RT-PCR, who had a fever at Baseline.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Oseltamivir (TAMIFLU®) 100 mg | Oseltamivir (TAMIFLU®) 200 mg | Oseltamivir Open Label
Number analyzed (Participants) | 7 | 6 | 2
Hours | 11.8 [7.8 to 43.5] | 18.6 [8.4 to 66.8] | 47.7 [NA to NA] — Data available for only 1 patient (1 patient was censored).

10. Secondary Outcome: Number of Participants With Viral Resistance
Description: Nasal and Throat swabs were collected on Days 1, 4, 6, 11, 15 and 30 and were sent to a central laboratory for testing. Viral resistance was determined by phenotypic and genotypic testing.
Time Frame: 30 days
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Oseltamivir (TAMIFLU®) 100 mg | Oseltamivir (TAMIFLU®) 200 mg | Oseltamivir Open Label
Number analyzed (Participants) | 30 | 32 | 10
Participants | 1 | 1 | 0

11. Secondary Outcome: Percentage of Participants With Influenza Symptoms
Description: Influenza (flu) symptoms were nasal congestion, sore throat, cough, aches and pains, fatigue, headache or chills.
Time Frame: Days 1, 11, 15, 30
Population: Intent-to-Treat population included all treated participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Oseltamivir (TAMIFLU®) 100 mg | Oseltamivir (TAMIFLU®) 200 mg | Oseltamivir Open Label
Number analyzed (Participants) | 49 | 50 | 14
Percentage of participants
  Day 1 | 100 | 100 | 93
  Day 11 | 63 | 64 | 79
  Day 15 | 51 | 44 | 64
  Day 30 | 33 | 26 | 64

ADVERSE EVENTS:
Description: Safety population included all participants who received treatment and had at least one post-treatment safety assessment. One patient in the 100 mg group actually received 200 mg and is included in the 200 mg group for safety.
Arm/Group | Oseltamivir (TAMIFLU®) 100 mg | Oseltamivir (TAMIFLU®) 200 mg | Oseltamivir Open Label
Serious Adverse Events (participants affected / at risk) | 9/48 | 5/51 | 7/14
Other Adverse Events (participants affected / at risk) | 17/48 | 18/51 | 10/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oseltamivir (TAMIFLU®) 100 mg (N=48) | Oseltamivir (TAMIFLU®) 200 mg (N=51) | Oseltamivir Open Label (N=14)
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 2 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lung infection pseudomonal (Infections and infestations) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oseltamivir (TAMIFLU®) 100 mg (N=48) | Oseltamivir (TAMIFLU®) 200 mg (N=51) | Oseltamivir Open Label (N=14)
Nausea (Gastrointestinal disorders) | 6 | 1 | 1
Vomiting (Gastrointestinal disorders) | 3 | 4 | 0
Constipation (Gastrointestinal disorders) | 2 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 4 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 4 | 1 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Infusion site pain (General disorders) | 3 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2
Hypertension (Vascular disorders) | 3 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.